CLINICAL TRIAL: NCT01078233
Title: Observational Safety Data Analysis From Routine Follow-up in the EuroSIDA Study of Patients Treated With Raltegravir in a Five-Year Post Authorization Period
Brief Title: Observational Data Analysis in EuroSIDA (MK-0518-058)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: EuroSIDA Coordinating Centre, Copenhagen HIV Programme (CHIP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0518-058; 2010_020 (Other: Merck); EP08025.005 (Other: Merck)
Record Dates: First submitted 2010-02-26; First posted 2010-03-02 (Estimated); Results first posted 2015-09-17 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: HIV-1 Infections
Keywords: HIV; antiretroviral treatment; HIV Cohort; Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Raltegravir Cohort: Participants with HIV-1 infection who started raltegravir on or after 21 December 2007 (the authorization date in the European Union) and had at least 1 month prospective follow-up in the Raltegravir Cohort. Participants from the Historical Cohort and Concurrent Cohort were eligible for inclusion in the Raltegravir Cohort.
- Historical Cohort: Participants with HIV-1 infection who started a new antiretroviral drug as part of a combination antiretroviral therapy (cART) regimen on or after 1 January 2006 and before 21 December 2007. Participants had no previous exposure to the new drug and had at least 1 month prospective follow-up in the Historical Cohort.
- Concurrent Cohort: Participants with HIV-1 infection who started a new antiretroviral drug other than raltegravir as part of a cART regimen on or after 21 December 2007. Participants had no previous exposure to the new drug and had at least 1 month prospective follow-up in the Concurrent Cohort. Participants from the Historical Cohort were eligible for inclusion in the Concurrent Cohort.

SUMMARY:
The main objective of the study is to monitor health outcomes associated with antiretroviral drugs in a population of HIV-infected patients.

DETAILED DESCRIPTION:
Time Perspective: Retrospective and Prospective

ELIGIBILITY:
Inclusion Criteria:

* Adults 16 years old and older with HIV-1

Exclusion Criteria:

* Subjects will be excluded if they have no prospective follow up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults 16 years old and older in the EuroSIDA database
Sampling Method: Non-Probability Sample
Enrollment: 6617 (Actual)
Dates: Start 2008-05-05 (Actual); Primary Completion 2014-03-06 (Actual); Study Completion 2014-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Cozzi-Lepri A, Zangerle R, Machala L, Zilmer K, Ristola M, Pradier C, Kirk O, Sambatakou H, Fatkenheuer G, Yust I, Schmid P, Gottfredsson M, Khromova I, Jilich D, Flisiak R, Smidt J, Rozentale B, Radoi R, Losso MH, Lundgren JD, Mocroft A; EuroSIDA Study Group. Incidence of cancer and overall risk of mortality in individuals treated with raltegravir-based and non-raltegravir-based combination antiretroviral therapy regimens. HIV Med. 2018 Feb;19(2):102-117. doi: 10.1111/hiv.12557. Epub 2017 Oct 6. PMID 28984429
- See also: EUPAS Register (EUPAS17912) — http://www.encepp.eu/encepp/viewResource.htm?id=18914
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0518-058&kw=0518-058&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The analyses in this study are based on data collected from a cohort of HIV-1-infected participants in a setting of routine clinical care in Europe (EuroSIDA Cohort Study). Participants could contribute data to more than one cohort, but no overlap in follow-up time was allowed.
Groups:
- Raltegravir Cohort Only: Participants with HIV-1 infection who started raltegravir on or after 21 December 2007 (the authorization date in the European Union). Participants had no previous exposure to the new drug and had at least 1 month prospective follow-up in this cohort. These participants contributed data only to the Raltegravir Cohort.
- Historical and Raltegravir Cohorts Only: Participants with HIV-1 infection who 1) started a new antiretroviral drug as part of a combination antiretroviral therapy (cART) regimen on or after 1 January 2006 and before 21 December 2007 and had at least 1 month prospective follow-up in the Historical Cohort, and 2) started raltegravir on or after 21 December 2007 and had at least 1 month prospective follow-up in the Raltegravir Cohort. These participants contributed data to the Historical Cohort and the Raltegravir Cohort.
- Historical Cohort Only: Participants with HIV-1 infection who started a new antiretroviral drug as part of a cART regimen on or after 1 January 2006 and before 21 December 2007 and had at least 1 month prospective follow-up in this cohort. These participants contributed data only to the Historical Cohort.
- Historical and Concurrent Cohorts: Participants with HIV-1 infection who 1) started a new antiretroviral drug as part of a cART regimen on or after 1 January 2006 and before 21 December 2007 and had at least 1 month prospective follow-up in the Historical Cohort, and 2) started a new antiretroviral drug other than raltegravir as part of a cART regimen on or after 21 December 2007, had no previous exposure to the new drug and had at least 1 month prospective follow-up in the Concurrent Cohort. These participants contributed data to the Historical Cohort and the Concurrent Cohort.
- Concurrent Cohort Only: Participants with HIV-1 infection who started a new antiretroviral drug other than raltegravir as part of a cART regimen on or after 21 December 2007, had no previous exposure to the new drug and had at least 1 month prospective follow-up in the Concurrent Cohort. These participants contributed data only to the Concurrent Cohort.
- Concurrent and Raltegravir Cohorts Only: Participants with HIV-1 infection who 1) started a new antiretroviral drug other than raltegravir as part of a cART regimen on or after 21 December 2007, had no previous exposure to the new drug and had at least 1 month prospective follow-up in the Concurrent Cohort, and 2) started raltegravir on or after 21 December 2007 and had at least 1 month prospective follow-up in the Raltegravir Cohort. These participants contributed data to the Concurrent Cohort and the Raltegravir Cohort.
Period: Overall Study
Arm/Group | Raltegravir Cohort Only | Historical and Raltegravir Cohorts Only | Historical Cohort Only | Historical and Concurrent Cohorts | Concurrent Cohort Only | Concurrent and Raltegravir Cohorts Only
Started | 656 | 296 | 1681 | 631 | 3199 | 154
Completed | 656 | 296 | 1681 | 631 | 3199 | 154
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir Cohort Only | Historical and Raltegravir Cohorts Only | Historical Cohort Only | Historical and Concurrent Cohorts | Concurrent Cohort Only | Concurrent and Raltegravir Cohorts Only | Total
Number analyzed (Participants) | 656 | 296 | 1681 | 631 | 3199 | 154 | 6617
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 49 [44 to 55] | 49 [44 to 55] | 44 [39 to 50] | 47 [41 to 53] | 42 [34 to 50] | 50 [45 to 57] | 44 [37 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 72 | 422 | 174 | 873 | 27 | 1744
  Male | 480 | 224 | 1259 | 457 | 2326 | 127 | 4873

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Malignancy
Description: All-type malignancy, including both Acquired Immune Deficiency Syndrome (AIDS)-defining and non-AIDS-defining malignancy, was evaluated. Only the first occurrence of any malignancy type was counted for each participant.
Time Frame: Historical Cohort: up to 24 months (January 2006 to December 2007); Raltegravir and Concurrent Cohorts: up to 68 months (December 2007 to July 2013)
Population: Intention-to-Treat analysis included follow-up until the end of the follow-up period for the cohort, regardless of whether or not raltegravir or other drugs were discontinued.
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years of follow-up
Units Other Than Participants: Person years of follow-up
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1150 | 2608 | 3984
Number analyzed (Person years of follow-up) | 2712 | 2895 | 10035
Events per 100 person-years of follow-up | 1.29 [0.93 to 1.80] | 1.17 [0.84 to 1.64] | 0.81 [0.65 to 1.00]

2. Primary Outcome: Incidence of Clinically Important Hepatic Events
Description: Clinically important hepatic events were defined as either 1) hepatic encephalopathy (stage III or IV), or 2) discontinuation of raltegravir use where liver toxicity was listed as the reason for discontinuation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years of follow-up
Units Other Than Participants: Person years of follow-up
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1150 | 2608 | 3984
Number analyzed (Person years of follow-up) | 2750 | 2891 | 10086
Events per 100 person-years of follow-up | 0.11 [0.04 to 0.34] | 0.90 [0.61 to 1.32] | 0.28 [0.19 to 0.40]

3. Primary Outcome: Incidence of Lipodystrophy
Description: Lipodystrophy events were defined as the first report for either 1) loss of fat from extremities, buttocks, or face, or 2) accumulation of fat in abdomen, neck, breasts, or other defined location.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years of follow-up
Units Other Than Participants: Person years of follow-up
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1150 | 2608 | 3984
Number analyzed (Person years of follow-up) | 2750 | 2893 | 10033
Events per 100 person-years of follow-up | 0.15 [0.05 to 0.39] | 1.04 [0.73 to 1.48] | 0.64 [0.50 to 0.81]

4. Primary Outcome: Incidence of All-Cause Mortality
Description: All participant deaths were recorded
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years of follow-up
Units Other Than Participants: Person years of follow-up
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Number analyzed (Participants) | 1150 | 2608 | 3984
Number analyzed (Person years of follow-up) | 2782 | 2913 | 10149
Events per 100 person-years of follow-up | 0.86 [0.58 to 1.29] | 1.27 [0.92 to 1.75] | 0.68 [0.54 to 0.86]

ADVERSE EVENTS:
Description: Per protocol, adverse events were not collected as part of the study database; therefore, none were collected and the number at risk is zero
Arm/Group | Raltegravir Cohort | Historical Cohort | Concurrent Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No